CLINICAL TRIAL: NCT04768907
Title: Early Access Program With MaaT013 in Steroid-refractory Acute Gastrointestinal Graft Versus Host Disease
Acronym: ATLAS
Status: Available | Type: Expanded Access
Sponsor: MaaT Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: MPOHEAP
Record Dates: First submitted 2021-02-22; First posted 2021-02-24 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Acute Graft Versus Host Disease in Intestine; Steroid Refractory GVHD

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: MaaT013

SUMMARY:
MaaT013 is still in clinical development phase and is not approved yet for marketing in any region. During the development program, MaaT Pharma has undertaken initial development with closely related product candidates, leading to the Phase II HERACLES study in which MaaT013 preliminary safety and efficacy were assessed in the context of steroid-resistant, gastrointestinal aGraft versus Host Disease (SR-GI-aGvHD). In addition, a pivotal Phase III study (ARES trial) is planned.

In the absence of medical options in patients with gastrointestinal acute GvHD refractory to multiple lines of treatment, this early access program has been implemented.

DETAILED DESCRIPTION:
Acute Graft-versus-Host Disease (aGvHD) is a serious and life-threatening disease that arises as a complication of allogeneic hematopoietic stem cell transplantation (allo-HSCT). At the onset of aGvHD, skin is the most frequently affected region (80% of patients) while GI tract or liver are involved in about 50% of patients (Martin 1990). aGvHD symptoms for the lower GI tract include watery diarrhea (≥500 mL), severe abdominal pain or bloody diarrhea (Ferrara 2009). While the incidence of severe GI-aGvHD has slightly decreased during the past decade, treatment remains unsuccessful in most cases (Gooley 2010, Castilla Llorente 2014), with a 2-months overall survival (OS) rate of 22% in steroid non-responsive or steroid refractory (SR) patients, non-responders to ruxolitinib (Jagasia 2020).

MaaT013 (pooled allogeneic fecal microbiota) is a live biotherapeutic product being developed by MaaT Pharma (Lyon, France) for the treatment of steroid-resistant, gastrointestinal aGvHD (SR-GI-aGvHD) adult patients with refractory, not eligible or who have failed second-line systemic therapy.

MaaT013 is still in clinical development phase and is not approved yet for marketing in any region. During the development program, MaaT Pharma has undertaken initial development with closely related product candidates, leading to the Phase II HERACLES study in which MaaT013 preliminary safety and efficacy were assessed in the context of SR-GI-aGvHD. In addition, a pivotal Phase III study (ARES trial) is planned

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18
* Grade III-IV gastro intestinal acute graft versus host disease with or without involvement of other organs:
* patients resistant to corticosteroid (CS) and resistant to one or multiple lines of treatments
* patients who cannot tolerate CS tapering, i.e., begin of CS at 2.0 mg/kg/d, demonstrate response, but show disease progress before a 50% decrease from the initial starting dose of CS is achieved.
* acute GVHD with overlap syndrome

Exclusion Criteria:

* Active uncontrolled infection
* Relapsed/persistent malignancy requiring rapid immune suppression withdrawal
* Current or past veno-occlusive disease or other uncontrolled complication
* Absolute neutrophil count <500/µL for 3 consecutive days. Use of growth factor supplementation is allowed
* Absolute platelet count < 10 000/µL. Use of platelet infusion is allowed
* Current or past evidence of toxic megacolon, bowel obstruction or gastrointestinal perforation
* Known allergy or intolerance to trehalose or maltodextrin
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (46):
- Austria (2):
  - University Clinic - State Hospital of Innsbruck, Innsbruck
  - Ordensklinikum Linz Elisabethinen, Linz
- Belgium (2):
  - Az Sint-Jan Brugge Av, Bruges
  - Hub - Institut Jules Bordet, Brussels
- Foothills Medical Centre, Calgary, Canada
- France (28):
  - Chu Amiens Picardie Site Sud, Amiens
  - Chu Angers, Angers
  - Chu Besancon, Besançon
  - Chu Morvan, Brest
  - Chu de Caen, Caen
  - Chu Grenoble, Grenoble
  - Chu de Lille, Lille
  - Chu Limoges, Limoges
  - MaaT Pharma, Lyon
  - Institut Paoli Calmettes, Marseille
  - Chu Montpellier - Hopital Saint Eloi, Montpellier
  - Chru Nancy, Nancy
  - Chu Nantes, Nantes
  - Chu de Nice - L'Archet 1, Nice
  - Aphp - Hopital Sant Antoine, Paris
  - Aphp - Hopital Necker, Paris
  - Chu Bordeaux - Hopital Haut-Leveque, Pessac
  - Hopital Haut Leveque, Pessac
  - Chu Lyon Sud, Pierre-Bénite
  - Chu La Miletrie, Poitiers
  - Chu de Rennes - Hopital Pontchaillou, Rennes
  - Chu Rouen, Rouen
  - Crlcc Henri Becquerel, Rouen
  - Chu St Etienne, Saint-Priest-en-Jarez
  - Chu Strasbourg - Hopital de Hautepierre, Strasbourg
  - Institut de Cancerologie de Strabsourg, Strasbourg
  - Iuct - Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (5):
  - Berlin University Medical Center - Charite Hospital, Berlin
  - University Hospital Essen, Essen
  - Saarlan University Medical Center, Homburg
  - University Hospital Mannheim, Mannheim
  - Ulm University Medical Center, Ulm
- Italy (5):
  - Aou Ospedali Riuniti, Ancona
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - Gemelli University Hospital, Roma
  - Aou Citta Della Salute E Della Scienza, Torino
  - Santa Maria Della Misericordia Hospital, Udine
- Spain (2):
  - Hospital General Universitario Morales Meseguer, Murcia
  - La Fe University Hospital, Valencia
- University Hospital of Geneva, Geneva, Switzerland